CLINICAL TRIAL: NCT00006436
Title: Short-Course EPOCH - Rituximab in Untreated CD-20+ HIV-Associated Lymphomas
Brief Title: EPOCH and Rituximab to Treat Non-Hodgkin's Lymphoma in Patients With HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Max Gordon, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010030; 01-C-0030; NCT00020384 (obsolete NCT alias)
Record Dates: First submitted 2000-11-03; First posted 2000-11-06 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma, AIDS-related; Lymphoma, Large B-Cell, Diffuse
Keywords: AIDS; Malignancy; Antiretroviral; Chemotherapy; Monoclonal
MeSH Terms: conditions — Lymphoma, AIDS-Related; Lymphoma, Large B-Cell, Diffuse; Acquired Immunodeficiency Syndrome; Neoplasms | interventions — Rituximab; Filgrastim; Etoposide; Prednisone; Vincristine; Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1-Combination Chemo and Biological Therapy (Experimental): Combination chemo and biological therapy
  Interventions: Biological: Rituximab; Biological: Filgrastim; Drug: EPOCH

INTERVENTIONS:
Biological: Rituximab — 2 doses of rituximab every cycle: first dose on Day 1 and 2nd dose on Day 5
  Other Names: Rituxan
Biological: Filgrastim — Filgrastim day 6 until absolute neutrophil count (ANC) reaches 5000 after the nadir, every cycle
  Other Names: Neupogen
Drug: EPOCH — combination chemotheray: EPOCH every 3 weeks for minimum of 3 cycles and max of 6 cycles
  Other Names: etoposide, prednisone, vincristine, cyclophosphamide and doxorubicin hydrochloride

SUMMARY:
Background:

* Human immunodeficiency virus (HIV)-infected patients have a weakened immune system, and chemotherapy, which is used to treat lymphoma, probably causes further damage to the immune system.
* Limiting the amount of immune damage due to chemotherapy might decrease the number of infections and the risk of developing cancer in the future in HIV-infected patients with non-Hodgkin's lymphoma.

Objectives:

* To determine whether reducing the total amount of chemotherapy using a specific combination of drugs called EPOCH-R (etoposide, doxorubicin, vincristine, cyclophosphamide and rituximab) will rid the body of lymphoma quickly while decreasing the risk of infections and future cancers.
* To determine whether the lymphoma will remain undetectable for at least one year if treatment is stopped one cycle after the patient enters remission.

Eligibility:

-Patients with non-Hodgkin's lymphoma and HIV infection 4 years of age and older who have not been treated previously with rituximab or cytotoxic chemotherapy.

Design:

* Patients receive EPOCH-R in 3-week treatment cycles for at least three and no more than six cycles.
* The lymphoma is evaluated using computed tomography (CT) and positron emission tomography (PET) scans at the end of treatment cycles 2 and 3. A bone marrow biopsy is repeated after cycle 2 if a biopsy was initially positive on screening for participation in the study.
* Anti-HIV therapy is stopped before chemotherapy begins and is restarted when EPOCH-R treatment ends.
* Patients are monitored for treatment response with blood tests and imaging scans at baseline, when treatment ends, 2 months after treatment ends and then every 3 to 6 months for a total of 24 months following chemotherapy.

DETAILED DESCRIPTION:
Background:

This is a study to investigate in a preliminary fashion the feasibility of short course chemotherapy to participants with HIV-associated non-Hodgkin's lymphoma (HIV-NHL).

This study will investigate if the paradigm for treatment can be successfully changed from a standard of 6 cycles to one cycle beyond complete remission with 6 total allowable cycles.

Objective:

To assess with 90 percent probability that at least 50 percent of participants treated with short-course EPOCH-R (etoposide, doxorubicin, vincristine, cyclophosphamide and rituximab) will be progression free at one year.

Eligibility:

Aggressive B-lymphocyte antigen CD20 (CD20) positive Diffuse large B cell lymphoma (DLBCL).

HIV+ serology.

All stages (I-IV) of disease.

Eastern Cooperative Oncology Group (ECOG) Performance status 0-4.

Non-Hodgkin's Lymphoma (NHL) previously untreated with cytotoxic chemotherapy.

Age greater than or equal to 18 years.

May not be pregnant or nursing.

May not have received previous rituximab.

Design:

Participants will be treated every three weeks with a combination of EPOCH and rituximab for one cycle beyond complete remission (CR)/complete response unconfirmed (CRu) by computed tomography (CT) scan of all detectable tumors for a minimum of three and maximum of six cycles. Following cycle 2, CT, positron emission tomography scans (PET), and bone marrow biopsies (if initially positive) will be performed.

At the conclusion of the study, we will estimate whether the number of cycles can be reduced using the paradigm. If the cumulative number of participants to relapse exceeds 25 percent by 6 months, the study will be closed.

Following the completion of chemotherapy, restaging will be performed 2 months following the end of treatment, then every 3 months for one year, every 6 months for one year, then every 12 months until relapse, death, or loss to follow up.

Antiretroviral therapy (ART) will be given concurrently with treatment regimen.

To study the effects of treatment approach on parameters of HIV disease, measurements of cluster of differentiation 4 (CD4) cells and viral loads will be made at baseline and at the completion of therapy, and then 2 months following the end of treatment, and then every 3-6 months for a total of 24 months following chemotherapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Aggressive B-lymphocyte antigen CD20 (CD20) positive Diffuse Large B-cell lymphoma confirmed by Laboratory of Pathology, National Cancer Institute (NCI). Note: Participants with aggressive B-cell lymphoma of the plasmablastic lymphoma sub-type who do not have surface CD20 expression, are also eligible.

Human immunodeficiency virus (HIV) + serology.

All stages (I-IV) of disease.

Eastern Cooperative Oncology Group (ECOG) Performance status 0-4

Non-Hodgkin's Lymphoma (NHL) previously untreated with cytotoxic chemotherapy; however, participants may be entered if they have had prior cyclophosphamide for an urgent problem at diagnosis (e.g., epidural cord compression, superior vena cava syndrome) and/or a single dose of intrathecal methotrexate (MTX) at the time of the pre-treatment diagnostic lumbar puncture

Age greater than or equal to 18 years

Laboratory tests (unless impairment due to respective organ involvement by tumor):

* Creatinine less than or equal to 1.5 mg/dl or creatinine clearance greater than or equal to 50 ml/min
* Bilirubin less than 2.0 mg/dl, or total bilirubin less than or equal to 4.5 mg/dl with direct fraction less than or equal to 0.3 mg/dl in participants for whom these abnormalities are felt to be due to protease inhibitor therapy
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3x upper limit of normal (ULN) (AST and ALT less than or equal to 6x ULN for participants on hyperalimentation for whom these abnormalities are felt to be due to the hyperalimentation)
* Absolute neutrophil count (ANC) greater than or equal to 1000/mm(3)
* Platelet greater than or equal to 75,000/mm(3) (unless impairment due to Immune thrombocytopenic purpura (ITP)

Ability of participant to provide informed consent.

EXCLUSION CRITERIA:

Previous rituximab

Pregnancy or nursing.

- Doxorubicin, etoposide, vincristine and cyclophosphamide are teratogenic and may be excreted in milk.

Current clinical heart failure or symptomatic ischemic heart disease.

Serious underlying medical condition or infection other than HIV that would contraindicate subcutaneous (SC)-rituximab, etoposide phosphate, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride (hydroxydaunorubicin (EPOCH-R).

* Examples include, but are not limited to:
* Severe Acquired immunodeficiency syndrome (AIDS)-related wasting
* Sever intractable diarrhea
* Active inadequately treated opportunistic infection of the central nervous system (CNS)
* Primary CNS lymphoma

Primary CNS lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2001-01-29 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2024-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Max Gordon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
  All large-scale genomic sequencing data will be shared with subscribers to database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol genomic data sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).
  Genomic data are made available via database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Kurtz DM, Scherer F, Jin MC, Soo J, Craig AFM, Esfahani MS, Chabon JJ, Stehr H, Liu CL, Tibshirani R, Maeda LS, Gupta NK, Khodadoust MS, Advani RH, Levy R, Newman AM, Duhrsen U, Huttmann A, Meignan M, Casasnovas RO, Westin JR, Roschewski M, Wilson WH, Gaidano G, Rossi D, Diehn M, Alizadeh AA. Circulating Tumor DNA Measurements As Early Outcome Predictors in Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2018 Oct 1;36(28):2845-2853. doi: 10.1200/JCO.2018.78.5246. Epub 2018 Aug 20. PMID 30125215
- [Derived] Dunleavy K, Pittaluga S, Shovlin M, Steinberg SM, Cole D, Grant C, Widemann B, Staudt LM, Jaffe ES, Little RF, Wilson WH. Low-intensity therapy in adults with Burkitt's lymphoma. N Engl J Med. 2013 Nov 14;369(20):1915-25. doi: 10.1056/NEJMoa1308392. PMID 24224624
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-C-0030.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1-Combination Chemo and Biological Therapy: Combination chemo and biological therapy
  Rituximab: 2 doses of rituximab every cycle: first dose on Day 1 and 2nd dose on Day 5
  Filgrastim: Filgrastim day 6 until absolute neutrophil count (ANC) reaches 5000 after the nadir, every cycle
  Etoposide, prednisone, vincristine, cyclophosphamide and doxorubicin hydrochloride (EPOCH): combination chemotherapy: EPOCH every 3 weeks for minimum of 3 cycles and max of 6 cycles
Period: Overall Study
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Started | 68
Completed | 65
Not Completed | 3
Not completed — Refused further treatment | 2
Not completed — Declined to participate (before treatment started) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 66
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.36 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 32
  White | 31
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: PFS is the time interval from study entry to documented evidence of disease progression or death due to any cause. Progression is defined according to the Cheson response criteria. Disease progression is defined as increase of 25% or more in the sum of the products of the longest perpendicular diameters of all measured lesions compared to the smallest previous measurements, or the appearance of any new lesion(s). Confidence intervals were made, and a Kaplan-Meier curve of progression free survival was constructed.
Time Frame: The participants were followed for a median of 15.4 years.
Population: One participant declined to participate before treatment started.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 67
years | 13.8 [10.2 to NA] — Upper end confidence interval is not estimable because the number of events beyond the median, and their timing, does not permit calculation of the upper confidence interval.

2. Primary Outcome: Progression Free Survival at 1 Year
Description: PFS is the time interval from start of treatment to documented evidence of disease progression. Progression is defined according to the Cheson response criteria. Disease progression as indicated by imaging scans at one year following therapy. Disease progression is defined as increase of 25% or more in the sum of the products of the longest perpendicular diameters of all measured lesions compared to the smallest previous measurements, or the appearance of any new lesion(s).
Time Frame: 1 year
Population: One participant declined to participate before treatment started.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 67
percentage of participants | 79.1 [67.3 to 87.1]

3. Secondary Outcome: Number of Participants With ≥ Grades 3-5 Non-hematologic Toxicity
Description: Non-hematologic (i.e., not begin in bone marrow or blood) toxicity was assessed by the Common Toxicity Criteria (CTC v2.0). Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to date off study, approximately 209 months and 17 days.
Population: One participant declined to participate before treatment started.
Measure: Count of Participants; unit: Participants
Groups:
- Grade 3: Grade 3 is serious.
- Grade 4: Grade 4 is life threatening.
- Grade 5: Grade 5 is death related to adverse event.
Arm/Group | Grade 3 | Grade 4 | Grade 5
Number analyzed (Participants) | 67 | 67 | 67
Participants
  Serious infection | 17 | 0 | 0
  Neurologic event | 0 | 0 | 0
  Syncope | 1 | 0 | 0
  Confusion | 1 | 0 | 0
  Motor neuropathy | 0 | 1 | 0
  Vision disturbance | 1 | 0 | 0
  Hyperglycemia | 4 | 0 | 0
  Hypophosphatemia | 2 | 1 | 0
  Hypocalcemia | 2 | 0 | 0
  Hypokalemia | 1 | 1 | 0
  Hyponatremia | 1 | 0 | 0
  Dehydration | 1 | 0 | 0
  Mucositis/Stomatitis | 6 | 0 | 0
  Liver test abnormalities | 6 | 1 | 0
  Pancreatitis | 1 | 0 | 0
  Diarrhea | 2 | 0 | 0
  Constipation | 1 | 0 | 0
  Serious hemorrhage | 5 | 1 | 0
  Fatigue | 2 | 0 | 0
  Headache | 5 | 0 | 0
  Bone pain | 1 | 0 | 0
  Nausea | 0 | 1 | 0
  Anorexia | 0 | 1 | 0
  Hypoxia | 0 | 4 | 1
  Myelodysplastic syndrome | 0 | 0 | 1

4. Secondary Outcome: Median Overall Survival
Description: Overall survival is time from treatment start date until date of death or date last known alive.
Time Frame: The participants were followed for survival for a median of 15.4 years.
Population: One participant declined to participate before treatment started.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 67
years | 14.2 [13.2 to NA] — Upper end confidence interval is not estimable because the number of events beyond the median, and their timing, does not permit calculation of the upper confidence interval.

5. Secondary Outcome: 1 Year Overall Survival
Description: Overall survival is time from treatment start date until date of death or date last known alive.
Time Frame: 1 year
Population: One participant declined to participate before treatment started.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 67
percentage of participants | 83.7 [71.0 to 91.2]

6. Secondary Outcome: Median Duration of Complete Response/Complete Response Unconfirmed
Description: Complete response (CR) was assessed by the Cheson response criteria. Complete response is disappearance of all signs and symptoms of lymphoma for a period of at least one month. All lymph nodes and nodal masses must have regressed to normal size (1.5 cm in their greatest transverse diameter for nodes > 1.5 cm before therapy).
  Complete response unconfirmed (CRu) is when a residual lymph node mass > 1.5 cm in greatest transverse diameter that has regressed by > 75% in sum of the products of the greatest diameters, does not change over the last two treatments, and any biopsies obtained are negative will be considered to be in CR. In organs involved by disease, any residual lesions that have decreased by > 75% in sum of the products of the greatest diameters or are < 1 cm, are consistent with scar, and stable over the last two treatments will be considered to fulfill criteria for CR.
Time Frame: The participants were followed for duration of complete response or complete response unconfirmed for a median of 15.4 years.
Population: One participant declined to participate before treatment started.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 67
years | 13.9 [13.1 to NA] — Upper end confidence interval is not estimable because the number of events beyond the median, and their timing, does not permit calculation of the upper confidence interval.

7. Secondary Outcome: Percentage of Participants With CR/CRu Lasting 1 Year
Description: as for outcome 6
Time Frame: 1 year
Population: One participant declined to participate before treatment started.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 67
percentage of participants | 82.5 [70.7 to 89.9]

8. Secondary Outcome: Number of Participants With at Least One Hematologic Toxicity Event of Febrile Neutropenia
Description: Toxicity was assessed by the Common Toxicity Criteria (CTC v2.0). Febrile neutropenia is defined as a life-threatening complication requiring hospitalization and urgent broad-spectrum antibiotics.
Time Frame: Date treatment consent signed to date off study, approximately 209 months and 17 days.
Population: One participant declined to participate before treatment started.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 67
Participants | 18

9. Secondary Outcome: Number of Cycles of Hematologic Toxicity
Description: Cumulative number of cycles of hematologic toxicity. Hematologic (i.e., decrease in bone marrow and blood cells) toxicity was assessed by the Common Toxicity Criteria (CTC v2.0).
Time Frame: Up to 112 cycles (each cycle is 21 days + 7 days window)
Population: One participant declined to participate before treatment started.
Measure: Number; unit: cycles
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 67
cycles
  Febrile neutropenia | 25
  Neutropenia with a Nadir <500 cells/mm^3 | 112
  Neutropenia with a Nadir <100 cells/mm^3 | 77
  Thrombocytopenia with a Nadir <50,000 platelets/mm^3 | 40
  Thrombocytopenia with a Nadir <25,000 platelets/mm^3 | 6
  Anemia: hemoglobin <8 g/dL | 36

10. Secondary Outcome: Overall Response
Description: Overall response was determined by the Cheson Response Criteria. Participants with either a complete response (CR), complete response unconfirmed or partial response were considered responders. Less than a partial response was considered a non-response to therapy (i.e., Stable Disease and/or Progressive Disease). Complete response was defined as the disappearance of all signs and symptoms of lymphoma for a period of at least one month. All lymph nodes and nodal masses must have regressed to normal size. Complete response unconfirmed is a residual lymph node mass > 1.5 cm in greatest transverse diameter that has regressed by > 75% in sum of the products of the greatest diameters, does not change over the last two treatments, and any biopsies obtained are negative will be considered to be in CR. Partial response is defined as a 50% or greater decrease in the sum of the products of the longest perpendicular diameters of all measured lesions lasting for a period of at least one month.
Time Frame: The participants were followed for an average of 6 months to determine response to therapy.
Population: One participant declined to participate before treatment started, and one participant was not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 66
Participants
  Complete Response | 53
  Complete Response Unconfirmed | 10
  Partial Response | 1
  Non-Responder - Stable Disease | 1
  Non-Responder - Progressive Disease | 1

11. Secondary Outcome: Percentage of Participants With Complete Response
Description: Complete response was assessed by the Cheson Response Criteria. Complete response is disappearance of all signs and symptoms of lymphoma for a period of at least one month. All lymph nodes and nodal masses must have regressed to normal size (1.5 cm in their greatest transverse diameter for nodes > 1.5 cm before therapy).
Time Frame: The participants were followed for an average of 6 months to determine response to therapy.
Population: One participant declined to participate before treatment started, and one participant was not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 66
percentage of participants | 95

12. Secondary Outcome: Median Interim Positron Emission Tomography (PET) Positive Progression Free Survival (PFS)
Description: PFS is the time interval from start of treatment to documented evidence of disease progression or death from any cause. Disease progression was assessed by positron emission tomography scans after 2 cycles (each cycle is 21 days + 7 days window) of therapy using the Deauville criteria. Deauville score of 4 or 5 is considered positive on interim PET scan while a Deauville score of 1 or 2 or 3 is considered negative. The outcomes of the Deauville score was compared to determine PET positive progression free survival.
Time Frame: Participants were followed for up to 10.2 years to determine their response on interim PET scans.
Population: 27 participants had no PET scan.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 41
years
  Interim PET positive participants: number analyzed (Participants) | 13
  Interim PET positive participants | 10.2 [0.4 to NA] — Upper end of the CI is not estimable because the number of events beyond the median, and their timing, does not permit calculation of the upper confidence interval.
  Interim PET negative participants: number analyzed (Participants) | 28
  Interim PET negative participants | NA [NA to NA] — Median not reached and confidence intervals cannot be reported because of the timing of the events relative to the follow-up of all participants.
Statistical Analysis 1: Comparison: Arm 1-Combination Chemo and Biological Therapy; Test type: Superiority; p = 0.10, Two-tailed log rank test; Compared the PFS of interim PET positive participants to the PFS of interim PET negative

13. Secondary Outcome: 1 Year Interim Positron Emission Tomography (PET) Positive Progression Free Survival (PFS)
Description: 1-year PFS is defined as participants who remain free of disease progression or death at one year from study entry. We compared the 1-year PFS of participants with negative results on interim positron emission tomography (PET) scans to those with positive results on interim PET scans.
  PFS is defined as the time interval from start of treatment to documented evidence of disease progression or death from any cause. Disease progression was assessed by positron emission tomography scans after 2 cycles of therapy using the Deauville criteria. Deauville score of 4 or 5 is considered positive on interim PET scan while a Deauville score of 1 or 2 or 3 is considered negative. The outcomes of the Deauville score was compared to determine PET positive progression free survival.
Time Frame: 1 year
Population: 27 participants had no PET scan.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 41
percentage of participants
  Interim PET scan positive 1-year PFS: number analyzed (Participants) | 13
  Interim PET scan positive 1-year PFS | 61.5 [30.8 to 81.8]
  Interim PET scan negative 1 year PFS: number analyzed (Participants) | 28
  Interim PET scan negative 1 year PFS | 89.3 [70.4 to 96.3]

14. Secondary Outcome: Recovery of CD4 T Cells (CD4) Counts
Description: Participants with human immunodeficiency virus (HIV) who undergo chemotherapy may have a delay in the recovery of their normal CD4+ T-cells. This delay could result in an increased risk of infection. Recovery of CD4 cells counts is the time from end of therapy until the time that the CD4 counts first reached above 200 cells/uL.
Time Frame: From the end of chemotherapy every 3 months for the first 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 67
months | 2.5 [0 to 24]

15. Secondary Outcome: Recovery of Human Immunodeficiency Virus (HIV) Viral Load
Description: The HIV viral load is a measure of actively replicating virus in the blood. If no anti-retroviral therapy is given, then reduction of this HIV viral load to manageable levels might risk infection. In our study, the recovery of HIV viral load was measured the time from the initiation of antiretroviral therapy until the viral load was undetectable or < 50 copies.
Time Frame: Either following or concurrently with combination chemo and biological therapy, approximately every 6 to 8 weeks after therapy was completed up to 16 months
Measure: Median (Full Range); unit: months
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 67
months | 2 [0 to 16]

16. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Toxicity Criteria (CTC v2.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Toxicity Criteria (CTC v2.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 209 months and 17 days.
Population: One participant declined to participate before treatment started.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
Number analyzed (Participants) | 67
Participants | 66

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 209 months and 17 days.
Description: One participant declined to participate before treatment started.
Arm/Group | Arm 1-Combination Chemo and Biological Therapy
All-Cause Mortality (participants affected / at risk) | 12/67
Serious Adverse Events (participants affected / at risk) | 23/67
Other Adverse Events (participants affected / at risk) | 66/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1-Combination Chemo and Biological Therapy (N=67)
Abdominal pain or cramping (General disorders) | 1 (1)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiovascular/Arrhythmia-Other (Asystole) (Cardiac disorders) | 1 (1)
CNS hemorrhage/bleeding (Nervous system disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Constitutional Symptoms-Other (Death- Accident/Overdose) (General disorders) | 1 (1)
Creatinine (Renal and urinary disorders) | 1 (2)
Dehydration (Gastrointestinal disorders) | 1 (1)
Edema (Cardiac disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 6 (9) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (Infections and infestations) | 3 (3)
Headache (Nervous system disorders) | 4 (4)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Gastrointestinal disorders) | 1 (1)
Hemorrhage-Other (alveolar) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypophosphatemia (metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Infection without neutropenia (Infections and infestations) | 3 (3)
Melena/GI bleeding (Gastrointestinal disorders) | 1 (1)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Neuropathy - motor (Nervous system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Other (Excludes metastasis from initial primary site: B-cell lymphoma) excludes metastasis from initial primary
Secondary Malignancy-Other (Myelodysplasia/Leukemia) excludes metastasis from initial primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Seizure(s) (Nervous system disorders) | 1 (1)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 2 (2)
Vision-photophobia (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1-Combination Chemo and Biological Therapy (N=67)
Abdominal pain or cramping (Gastrointestinal disorders) | 10 (10)
Alkaline phosphatase (Hepatobiliary disorders) | 22 (34)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 9 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (28)
Amylase (Metabolism and nutrition disorders) | 3 (5)
Anorexia (Gastrointestinal disorders) | 17 (23)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 4 (5)
Bicarbonate (Metabolism and nutrition disorders) | 8 (9)
Bilirubin (Hepatobiliary disorders) | 16 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 30 (44)
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiovascular/Arrhythmia-Other (Tachycardia) (Cardiac disorders) | 1 (1)
Chest pain (non-cardiac and non-pleuritic) (Musculoskeletal and connective tissue disorders) | 7 (8)
Confusion (Nervous system disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 25 (38)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (19)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 3 (3)
Creatinine (Renal and urinary disorders) | 6 (7)
Dehydration (Gastrointestinal disorders) | 5 (7)
Dermatology/Skin-Other (BACTBRABAN) (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin-Other (Blisters on hands & feet) (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin-Other (Left leg erythema) (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin-Other (Erythema derm other) (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 28 (45)
Dizziness/lightheadedness (Nervous system disorders) | 9 (11)
Dry eye (Endocrine disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspepsia/heartburn (Gastrointestinal disorders) | 5 (6)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 14 (17)
Dysuria (painful urination) (Renal and urinary disorders) | 1 (1)
Earache (otalgia) (Ear and labyrinth disorders) | 1 (1)
Edema (Cardiac disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Erectile impotence (Reproductive system and breast disorders) | 1 (1)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 32 (57)
Febrile neutropenia (Infections and infestations) | 17 (21) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 14 (18)
Flatulence (Gastrointestinal disorders) | 5 (6)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Gastrointestinal-Other (Appendicitis-Appendectomy performed) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal-Other (Fecal incontinence) (Gastrointestinal disorders) | 1 (1)
Hallucinations (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 30 (47)
Hematemesis (Gastrointestinal disorders) | 1 (1)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 60 (157)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Gastrointestinal disorders) | 2 (2)
Hemorrhage-Other (Hemorrhage, GI) (Gastrointestinal disorders) | 1 (1)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 29 (50)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (5)
Hypermagnesemia (Metabolism and nutrition disorders) | 8 (9)
Hypernatremia (Metabolism and nutrition disorders) | 4 (4)
Hypertension (Cardiac disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 5 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 25 (35)
Hypocalcemia (Metabolism and nutrition disorders) | 25 (31)
Hypoglycemia (Metabolism and nutrition disorders) | 6 (8)
Hypokalemia (Metabolism and nutrition disorders) | 16 (27)
Hypomagnesemia (Metabolism and nutrition disorders) | 27 (44)
Hyponatremia (Metabolism and nutrition disorders) | 25 (41)
Hypophosphatemia (Metabolism and nutrition disorders) | 14 (17)
Hypotension (Cardiac disorders) | 7 (9)
Hypothyroidism (Endocrine disorders) | 1 (1)
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 2 (2)
Infection (Infections and infestations) | 19 (26) — (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e9/L)
Infection without neutropenia (Infections and infestations) | 21 (39)
Infection/Febrile Neutropenia-Other (Infection with Grade 2 neutropenia) (Infections and infestations) | 1 (1)
Inner ear/hearing (Ear and labyrinth disorders) | 1 (1)
Insomnia (Nervous system disorders) | 10 (13)
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 61 (193)
Lipase (Metabolism and nutrition disorders) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 58 (169)
Memory loss (Nervous system disorders) | 1 (1)
Mood alteration-anxiety, agitation (Nervous system disorders) | 3 (6)
Mood alteration-depression (Nervous system disorders) | 8 (10)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 5 (7)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 14 (15)
Nail changes (Skin and subcutaneous tissue disorders) | 5 (9)
Nausea (Gastrointestinal disorders) | 33 (62)
Neuropathic pain (Nervous system disorders) | 2 (4) — (e.g., jaw pain, neurologic pain, phantom limb pain, post-infectious neuralgia, or painful neuropathies)
Neuropathy-sensory (Nervous system disorders) | 31 (54)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 62 (178)
Pain-Other (Back pain) (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain-Other (Neck pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Other (Pain -Other (sacral)) (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain-Other (Pain - Other (lower back)) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Other (Tooth pain) (Gastrointestinal disorders) | 1 (1)
Pain-Other (Myositis) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Other (Left leg pain_) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Other (bone marrow (BM) biopsy site) (General disorders) | 1 (1)
Pain-Other (pain behind eye) (Eye disorders) | 1 (1)
Pain-Other (Pain at port site) (General disorders) | 1 (1)
Pain-Other (Right hip hematoma) (General disorders) | 1 (1)
Pain-Other (Epigastric pain) (Gastrointestinal disorders) | 1 (1)
Pain-Other (Leg and back pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Other (Back) (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain-Other (Generalized) (General disorders) | 1 (1)
Pain-Other (Tooth abscess) (Gastrointestinal disorders) | 1 (1)
Pain-Other (Mild left side plank pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Partial thromboplastin time (PTT) (Investigations) | 10 (11)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 3 (4)
Platelets (Blood and lymphatic system disorders) | 56 (138)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Proctitis (Gastrointestinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Prothrombin time (PT) (Investigations) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9 (11)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 3 (3)
Rectal or perirectal pain (proctalgia) (Gastrointestinal disorders) | 4 (4)
Renal/Genitourinary-Other (Vaginal blisters) (Renal and urinary disorders) | 1 (1)
Rigors, chills (General disorders) | 6 (7)
Seizure(s) (Nervous system disorders) | 1 (1)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 31 (54)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 33 (62)
Sinus tachycardia (Cardiac disorders) | 6 (7)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 36 (61)
Sweating (diaphoresis) (General disorders) | 6 (6)
Syncope (fainting) (Nervous system disorders) | 2 (2)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 12 (16)
Tearing (watery eyes) (Eye disorders) | 2 (2)
Thrombosis/embolism (Cardiac disorders) | 5 (5)
Transfusion: Platelets (Blood and lymphatic system disorders) | 12 (48)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 25 (69)
Tumor lysis syndrome (Renal and urinary disorders) | 1 (1)
Tumor pain (onset or exacerbation of tumor pain due to treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 5 (5)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 4 (4)
Vision-flashing lights/floaters (Eye disorders) | 1 (1)
Vision-photophobia (Eye disorders) | 4 (4)
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 28 (44)
Weight gain (General disorders) | 1 (1)
Weight loss (General disorders) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT00006436/Prot_SAP_003.pdf
  • Informed Consent Form (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT00006436/ICF_001.pdf